CLINICAL TRIAL: NCT07136545
Title: A Phase I/II Trial of HCB101 in Combination With Pembrolizumab for Patients With Platinum-Refractory, Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (SirH&N Trial)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: FBD Biologics Limited (Industry); National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Mu-Hsin Chang, Attending Physician, Taipei Veterans General Hospital, Taiwan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01-015B
Record Dates: First submitted 2025-08-05; First posted 2025-08-22 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCB101+Pembrolizumab (Experimental)
  Interventions: Drug: HCB101; Drug: Pembrolizumab

INTERVENTIONS:
Drug: HCB101 — QW
Drug: Pembrolizumab — 200 mg IV on Day 1, cycled every 21 days;

SUMMARY:
This is a non-randomized, open-label, dose-escalation and dose-expansion phase I/II clinical study to evaluate the safety, tolerability, and efficacy of HCB101 in combination with pembrolizumab in patients with platinum-refractory recurrent/metastatic HNSCC. The trial consists of two phases: the dose-escalation phase (I) and the dose-expansion phase (II).

Subjects will receive a weekly single dose of HCB101 IV infusion over 60 (±10) minutes on Days 1, 8, and 15 in each 21-day cycle in combination with pembrolizumab (200 mg IV day 1; given every 21 days) until unacceptable AE(s), radiographic or clinically documented disease progression, withdrawal of consent, loss to follow-up, death, or termination of the study whichever occurs first.

ELIGIBILITY:
* Inclusion Criteria

  * 1. Subjects are able to understand and willing to provide signed informed consent as described in protocol, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, including study visits and study-related procedures.
  * 2. Male and female subjects of ≥18 years of age, inclusive, at the time of signing the informed consent.
  * 3. With histologically/cytologically confirmed diagnosis of HNSCC
  * 4. With progression after 1st cisplatin based therapy for R/M HNSCC or within 6 months after cisplatin based CCRT
  * 5. Must have at least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
  * 6. Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at Screening.
  * 7. Have a life expectancy of ≥12 weeks (according to the Investigator's judgment).
  * 8. Have adequate organ function, as indicated by the following laboratory parameters in below (had not received a blood transfusion, apheresis infusion, erythropoietin, granulocyte colony-stimulating factor, and other relevant medical support within 14 days prior to the administration of the first dose of study intervention).

    * a) Absolute neutrophil count ≥1.5 × 109/L
    * b) Platelets ≥75 × 109/L
    * c) Hemoglobin ≥9.5 g/dL
    * d) Total bilirubin ≤1.5 × upper limit of normal (ULN), <3.0 × ULN if known Gilbert's disease
    * e) Alanine aminotransferase and aspartate aminotransferase ≤3× ULN and ≤5× ULN for subject with liver metastasis
    * f) Creatinine clearance ≥50 mL/min (using Cockcroft Gault equation)
    * g) Coagulation: International normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (aPTT) ≤1.5× ULN (The INR applies only to subjects who do not receive therapeutic anticoagulation). For subjects receiving therapeutic anticoagulation, the INR should be within the therapeutic range for the intended use of the anticoagulants.)
  * 9. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test during the Screening Period (within 7 days prior to the first dose of the study intervention).
* Exclusion Criteria

  * 1. Medical Conditions:

    * a) With a known history of hypersensitivity to any components of the study intervention.
    * b) Subjects who have other malignancies requiring treatment within 2 years prior to the first dose of study intervention will be excluded, except for radically treated locally curable basal or squamous cell skin cancer and other malignancies that have been treated with no relapse within 2 years.
    * c) Primary tumor in the central nervous system (CNS), or active or untreated CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate, provided they are clinically stable for at least 28 days and have no evidence of new or enlarging brain metastases and no requirements for high-dose corticosteroids 14 days prior to dosing with study intervention. Subjects on low-dose corticosteroids (<20 mg prednisolone or equivalent per day) may participate.
    * d) Clinically significant cardiovascular condition, including 1)History of congestive heart failure (New York Heart Association Class >2), with only heart failure with preserved ejection fraction (HFpEF) included; 2)History of unstable angina within 6 months prior to the first dose of study intervention; 3)New-onset angina or myocardial infarction within 6 months prior to the first dose of study intervention; 4)New-onset of atrial fibrillation, supraventricular arrhythmia, or ventricular arrhythmia within 6 months prior to the first dose of study intervention and still in unstable condition and requiring treatment or intervention. History of atrial fibrillation, supraventricular arrhythmia, or ventricular arrhythmia will be allowed, provided the condition is stably controlled.
    * e) History or presence of an abnormal ECG that, in the Investigator's opinion, is clinically meaningful (including QT interval corrected for heart rate using Fridericia's correction [QTcF] >470 msec at Screening, pacemaker installation, or previous diagnosis of congenital long QT syndrome).
    * f) Any previous treatment-related toxicities which have not recovered to ≤ Grade 1 as evaluated by National Cancer Institute, Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 or baseline, except alopecia and anemia (Note: subjects with chronic Grade 2 toxicities which are well managed and stable may be eligible per the discretion of the Investigator, Grade 2 chemotherapy-induced neuropathy.)
    * g) With known inherited or acquired bleeding disorders or bleeding diathesis.
    * h) With a previously documented diagnosis of hemolytic anemia or Evans Syndrome in the last 3 months.
    * i) With active autoimmune diseases that required systemic treatment (e.g., disease-modifying agents, corticosteroids, or immunosuppressants) within the past two years are excluded. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) is allowed.
    * j) With a history of or current non-infectious pneumonitis.
    * k) With a history of severe hypersensitivity to monoclonal antibodies.
  * 2. Prior/Concomitant Therapy/Treatment

    * a) Subjects who have undergone major surgery or radical radiotherapy within 28 days prior to the first dose of study intervention.
    * b) Subjects who have undergone any investigational or approved systemic cancer therapy (including chemotherapy, immunotherapy, hormonal therapy, and herbal/alternative therapies with anti-cancer indications or targeted therapy) within 14 days or 5 half lives, whichever is longer, prior to the first dose of the study intervention.
    * c) Subjects who have used herbal medication within 14 days prior to the first dose of the study intervention.
    * d) Subjects who are active using of vitamin K antagonist anticoagulant like warfarin. Use of low molecular weight heparin and factor Xa inhibitors will be permitted on a case-by-case basis. There will be no restriction for daily aspirin ≤ 100 mg/QD.
    * e) Subjects who have received any treatment targeting the CD47 or SIRPα pathway.
    * f) Subjects who have previously received pembrolizumab treatment.
    * g) Subjects who have received a live vaccine within 30 days prior to pembrolizumab administration.
    * h) Subjects diagnosed with immunodeficiency, receiving systemic steroid therapy, or having received any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab.
  * 3. Participation in another clinical study with an investigational product administered in the last 14 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study intervention. An investigational device was used within 28 days prior to the first dose of study intervention.
  * 4. Reproductive and breastfeeding

    * a) Women of reproductive potential who are unable to use effective contraception during treatment and for 4 months after the last dose.
    * b) Women who are breastfeeding during treatment and for 4 months after the last dose.
  * 5. Infections:

    * a) An uncontrolled acute infection, an active infection requiring systemic treatment, or subjects who have received systemic antibiotics within 7 days prior to the first dose of the study intervention (Note: prophylaxis use of systemic antibiotics treatment for upper tract infection is allowed as long as there is no violation of the requirement of concomitant medications).
    * b) Known history of human immunodeficiency virus (HIV) infection.
    * c) Active tuberculosis.
    * d) Known history of hepatitis B or hepatitis C infection. Subjects who test positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody.
  * 6. Any other medical (e.g., Child-Pugh class B or C, pulmonary, metabolic, congenital, endocrinal or CNS disease, etc.), psychiatric, or social condition deemed by the Investigator to be likely to interfere with a subject's rights, safety, welfare or ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with MTD of HCB101 in combination with pembrolizumab | 2 Years
  To evaluate the safety and efficacy of HCB101 in combination with pembrolizumab
Overall Rate Response (ORR) | 2 Years
  To evaluate the safety and efficacy of HCB101 in combination with pembrolizumab

SECONDARY OUTCOMES:
Number/incidence and percentage of subjects with AEs, SAEs, and TEAEs | 2 Years
  To characterize the safety profiles of HCB101 in combination with pembrolizumab.
Progression-Free Survival (PFS) | 2 Years
  To evaluate the anti-tumor activity of HCB101 in combination with pembrolizumab.
Quality of life (EORTC QLQ-H&N35) change | 2 Years
  To evaluate the quality of life (QOL) change after treatment of HCB101 in combination with pembrolizumab

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Hsin Chang, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (3):
- Taiwan (3):
  - Chang-Gung Memorial Hospital(Lin-Kou), Taoyuan District, Guishan District
  - National Taiwan University Hospital, Taipei, Taipei city
  - Taipei Veterans General Hospital, Taipei, taipei city

IPD SHARING:
Plan to Share IPD: Undecided